CLINICAL TRIAL: NCT03389087
Title: Single Arm, Exploratory and Open Phase II Clinical Trial of Apatinib Plus Etoposide Capsule as the Therapy of Advanced Small Cell Lung Cancer
Brief Title: Study of Apatinib Plus Etoposide Capsule as the Therapy of Advanced Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP053
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib and Etoposide Capsule (Experimental): Apatinib and Etoposide Capsule
  Interventions: Drug: Apatinib and Etoposide Capsule

INTERVENTIONS:
Drug: Apatinib and Etoposide Capsule — Apatinib 250mg/qd，po, A course of treatment need 28 days. Etoposide Capsule 25mg/d，po, from day 1-day 21.

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Apatinib Plus Etoposide Capsule as the Therapy of Advanced Small Cell Lung Cancer.

DETAILED DESCRIPTION:
Small cell lung cancer is a very aggressive cancer, often accompanied by distant metastases, with a poor prognosis. 5-year survival rate of less than 5%, untreated patients with an average survival of only 2-4 months. The investigators consider to add apatinib,a tyrosine kinase inhibitor of VEGF,to the therapy of these patients. The investigators designed the study to explore the possibility of apatinib Plus Etoposide Capsule as the Therapy of Advanced Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of small cell lung cancer.
2. ≥ 18 and ≤ 75 years of age.
3. According to RESCIST1.1 standard, there are evaluable target lesions.
4. Has received second-line standard treatment of recurrent or metastatic extensive stage small cell lung cancer.
5. Life expectancy of more than 3 months.
6. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 2.
7. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥ 1.5×109/L, PLT ≥ 100×109/L, HB ≥ 90 g/L, TBIL ≤ 1.5×ULN, ALT or AST ≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1.25×ULN, Cr clearance ≥ 45 mL/min.
8. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 6 months after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 6 months after last dose of study drug.
9. Signed the informed consent form prior to patient entry.

Exclusion Criteria:

1. Active brain metastases, meningococcal meningitis, patients with spinal cord compression, or imaging at CT or MRI examination revealed brain or pia mater disease（Patients who have completed treatment and whose symptoms are stable in the first 21 days of randomization may be enrolled in the study but may be diagnosed as having no intracerebral hemorrhage by MRI, CT or venography）；
2. Imaging (CT or MRI) showed that the tumor lesions were ≤ 5 mm from the major vessels or there was a central tumor invading local macrovascular；
3. Imaging (CT or MRI) showed significant cavitary or necrotic lung tumors, uncontrollable hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg, despite optimal medical therapy), grade II The above myocardial ischemia or myocardial infarction, poor control of arrhythmia (including QTc interval male ≥ 450 ms, female ≥ 470 ms); NYHA standards, Ⅲ ~ Ⅳ grade cardiac insufficiency, or cardiac ultrasound examination prompted left ventricular ejection Score (LVEF) <50%；
4. Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment；Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or the like；
5. Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above；
6. Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc.
7. Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (Including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening（Such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism and so on）；
8. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g；
9. Previously used anti-angiogenic drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No